CLINICAL TRIAL: NCT04281251
Title: Endoscopic Retrograde Appendicitis Therapy - a Pilot Study
Brief Title: Endoscopic Retrograde Appendicitis Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Associate Consultant, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2020.011
Record Dates: First submitted 2020-02-20; First posted 2020-02-24 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Acute Appendicitis
Keywords: appendicitis; endoscopic drainage
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: Single arm case series
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ERAT arm (Experimental): This is the treatment arm where endoscopic therapy of acute appendicitis would be performed
  Interventions: Procedure: Endoscopic retrograde appendicitis therapy

INTERVENTIONS:
Procedure: Endoscopic retrograde appendicitis therapy — Colonoscopy would be introduced until visualization of the appendiceal orifice. Catheter would be placed in the appendix and decompression performed. After removal of appendicolith, plastic stent would be placed for drainage of appendix.
  For patients successfully treated with initial endoscopic drainage, they would be re-admitted at 1 weeks after index procedure for repeat colonoscopy. After reaching the appendiceal orifice, the previous plastic stent would be removed. A contrast appendicogram would be repeated by introducing a wire-guided catheter in the appendix, and any residual fecalith would be removed. Finally, a repeat contrast appendicogram would be performed to confirm complete clearance of fecalith.

SUMMARY:
This is a prospective pilot study on the efficacy of endoscopic therapy for adult uncomplicated acute appendicitis. In recent years, antibiotics treatment has been a new alternative approach to surgical appendicectomy for acute appendicitis, however, there is a risk of failed antibiotics treatment and chance of recurrent appendicitis.

Endoscopic therapy of acute appendicitis (ERAT) has been recently described that involves colonoscopic insertion of plastic stent and removal of appendicolith. The investigators conduct this pilot study to investigate the feasibility, technical and clinical success rate of endoscopic retrograde appendicitis therapy among adult patients with uncomplicated acute appendicitis. 20 patients would be recruited for the pilot study.

DETAILED DESCRIPTION:
Acute appendicitis is one of the most common surgical emergencies in adult patients. The lifetime risk of developing acute appendicitis in the United States is 8.6% for males and 6.7% for females. For many decades, surgical appendicectomy is the gold standard of treatment of acute appendicitis. Appendicectomy could be performed in an open manner via a right lower abdominal incision, or more popular nowadays with the laparoscopic approach by placing three abdominal trocars. Earlier studies have identified high treatment success rate with both open and laparoscopic approaches, but adverse events were lower in laparoscopic group. Intra-abdominal abscesses were a potential concern with laparoscopic appendicectomy. In recent few years, antibiotics treatment for acute appendicitis has been a promising management option. By avoid the need of surgery and general anaesthesia, the non-operative approach was associated with a lower morbidity than the surgical approach. The major drawback of antibiotic treatment was the risk of failed primary treatment and subsequent recurrent appendicitis. A recent randomized controlled study demonstrated a primary clinical success treatment at index attack of 94.2%. 72.7% of the patients who received antibiotics alone did not require appendicectomy at 1-year follow-up. While antibiotics therapy could be a safe alternative to surgical therapy, many are still skeptical of the treatment due to the potential high recurrence rate.

Endoscopic therapy of acute appendicitis (Endoscopic retrograde appendicitis therapy, ERAT) was recently described recently in the literature. The technique involves a two-staged procedure with endoscopic plastic stent drainage of appendiceal orifice followed by stent and appendicolith retrieval. These were small case series conducted in China demonstrating technical feasibility and initial clinical success rate of this alternative approach. The technique has not been practiced in most centers across the world. The merit of endoscopic treatment lies in its potential to remove the appendicolith thereby reducing the recurrence rate. It could provide an invaluable treatment option that overcomes the drawback of high recurrence rate with antibiotics alone.

Given that the novel endoscopic technique has not been widely adopted, the investigators plan to conduct this pilot study to investigate the feasibility, technical and clinical success rate of endoscopic retrograde appendicitis therapy among adult patients with uncomplicated acute appendicitis.

ELIGIBILITY:
Inclusion criteria

1. Adult patients emergency admitted for suspected acute appendicitis
2. Age 18 - 70
3. Computed Tomography of the abdomen with contrast confirmed uncomplicated appendicitis, as evidenced by presence of a dilated, thickened wall appendix without perforation, abscess or gangrene.

Exclusion criteria

1. History of previous appendicitis
2. Evidence of perforation, abscess or gangrene of appendix on CT scan
3. Significant paralytic ileus as evidenced by dilated bowel loops on imaging
4. Evidence of co-existing acute surgical pathologies on the CT scan
5. Allergic to bowel preparation solution (Polyethylene glycol)
6. Marked electrolyte abnormalities, significant renal impairment (CrCl <30ml/min)
7. Coagulopathy (INR >1.5, platelet <50)
8. Pregnancy, or contraindication to fluoroscopy
9. Other cases deemed by the examining physician as unsuitable for safe treatment
10. Refusal to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical success rate | 30 days
  defined as completion of both endoscopic procedures without need for surgery or complications related to acute appendicitis

SECONDARY OUTCOMES:
Technical success rate | 30 days
  defined as successful completion of both endoscopic procedures
Rate of recurrent acute appendicitis, up to 1 year of index attack | 1 year
  defined as recurrent diagnosis of acute appendicitis
Rate of adverse events related to endoscopic procedures | 30 days
  Rate of adverse events, graded according to Common Terminology Criteria for Adverse Events.
Scale of post-operative pain | 7 days
  Graded by Visual Analogue Scale from 0-10, (10 being the most painful) from Day 1 to 7

CONTACTS AND LOCATIONS:
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No